CLINICAL TRIAL: NCT00364455
Title: Randomized Trial of Epoetin Alfa in Men With Hormone-refractory Prostate Cancer and Anemia.
Brief Title: Impact of Erythropoietin Treatment Versus Placebo on Quality-of-life in Patients With Advanced Prostate Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Ortho Inc., Canada (Industry)
Collaborators: Ontario Clinical Oncology Group (OCOG) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006118
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Prostate; Carcinoma
Keywords: Hormone refractory prostate cancer; Anemia; Quality-of-life
MeSH Terms: conditions — Carcinoma; Anemia | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of this study was to evaluate the effect of treatment with epoetin alfa (recombinant human erythropoietin) or placebo on anemia related quality-of-life and anemia in hormone-refractory (not responding to hormone therapy) prostate cancer patients.

DETAILED DESCRIPTION:
Anemia is a common problem experienced by patients with malignancy. Although cancer treatment such as systemic chemotherapy is an obvious cause, many cancer patients are anemic at presentation. Estimates in prostate cancer patients suggest that nearly 40% present with hemoglobin levels less than 120 g/L. The most common clinical manifestation of anemia is fatigue, although vertigo, loss of appetite, poor concentration and dyspnea (shortness of breath) can also occur. Anemia often leads to impairment of physical capacity, lowers patients' subjective sense of well-being, and diminishes their overall quality-of-life (QoL). The use of recombinant erythropoietin for patients with chronic anemia of end stage renal disease, acquired immune deficiency syndrome, or anemia of chronic disease in the setting of malignancy (cancer) is well established to provide benefit in reducing transfusion requirements. There exists a number of published data on QoL in cancer patients. Abels et al. published in 1991 initial results of clinical reports that specifically reported on QoL outcomes. The study actually consisted of a series of three concurrent randomized, double blind, placebo controlled trials conducted on groups of patients with a variety of underlying malignancies. The three studies included 124 patients not previously treated with systemic therapy, 132 patients treated systemically with cisplatinum containing chemotherapy regimens and 157 patients treated with non-cisplatinum containing regimens respectively. All patients had pre-treatment hemoglobins of less than 105 g/L or hematocrits (percentage of red blood cells in blood) of less than 32%. In each trial, patients randomized to receive recombinant erythropoietin had significantly greater increases in hematocrit than placebo patients. QoL parameters (as measured on a visual analog scale) were significantly improved in patients receiving erythropoietin who demonstrated an increase in hematocrit throughout the three studies. Overall QoL improved significantly over baseline, although individual studies only demonstrated a trend towards improvement. Littlewood et al. published in 2001 the results of a double-blind, placebo controlled multi-center study of 375 cancer patients receiving non-platinum containing chemotherapy. A baseline hemoglobin of less than or equal to 105 g/L, or a drop of 20 g/L with chemotherapy was required for eligibility. Patients were randomized 1:2 to either placebo or epoetin alfa, for up to 4 weeks following chemotherapy. Active treatment demonstrated significant effectiveness in increasing hemoglobin levels and reducing transfusion requirements. Significant improvement in all primary cancer- and anemia-specific QoL domains favoured epoetin alfa. Although clinical evidence suggests benefit beyond reduced transfusion requirements, many studies looking at impact on QoL have been uncontrolled by design, with variable quality and collection of QoL data. Since they have also involved patients with a myriad of primary malignancies, and previous therapies, the translation of results to site and situation specific clinical practice has been difficult. As erythropoiesis is a complex process that depends on inhibiting or stimulating cytokines, which may be regulated differently among various neoplastic diseases (i.e. different tumour types), studies in more homogenous groups of patients were deemed necessary to evaluate impact on QoL. Prostate cancer is the most common serious cancer in men. Despite advances in screening and treatment, progression to the incurable metastatic phase of the disease remains common. Androgen ablation therapy using surgery or drugs remains the standard of treatment, but inevitably, androgen resistance develops. Hormone refractory prostate cancer represents a spectrum of disease ranging from asymptomatic patients with only biochemical evidence of androgen resistance to end-stage disease characterized by extensive bone metastases, pain, wasting, reduced QoL, and a median survival of less than one year. Treatment of hormone refractory prostate cancer does not prolong survival, but may improve symptoms and QoL. Anemia is common in this group of patients, with hemoglobin levels of less than 120 g/L often seen (in up to 40% patients). Patients are also genrally older, often have co-morbid conditions, and transfusions for palliation are frequently given. A randomized, placebo-controlled study evaluating an intervention with epoetin alfa that could significantly improve QoL was thus carried out in hormone refractory prostate cancer patients. It was deemed that such an intervention, if successful, could have the potential to change current clinical practice. Moreover, improved QoL, in response to increased Hb levels, could also lead to a reduction in hospital admissions and to fewer transfusions in this patient population.

Patients were to receive either 40,000 IU epoetin alfa weekly or matching placebo subcutaneously for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological confirmed adenocarcinoma of the prostate or patients who have metastatic carcinoma of presumptive prostate origin as manifest by the presence of sclerotic bony metastases and a serum PSA level greater than the upper limit of normal
* Hemoglobin level at or below 120 g/L
* ECOG (Eastern Cooperative Oncology Group) Performance status of 0-2.

Exclusion Criteria:

* No known or suspected CNS metastasis (Cancer that has spread from the original (primary) tumor to the central nervous system)
* No other active concurrent malignancy, other than the underlying prostate cancer which is expected to influence QoL
* No blood transfusions within the last 14 days and no previous use of erythropoietin (i.e., that would impact baseline Hb)
* No anemia due to factors other than cancer/radiotherapy (i.e., hemolysis or gastrointestinal bleeding, evidence of untreated folate or vitamin B12 deficiency)
* No history of uncontrolled hypertension or diastolic blood pressure greater than 100 mmHg
* No mental incompetence, including psychiatric or addictive disorders which would preclude meaningful completion of quality-of-life questionnaires.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2002-12; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome was change in Quality of Life (FACT-An Anemia scale) from baseline to 16 weeks.

SECONDARY OUTCOMES:
QoL was measured at baseline, 4, 8, 12, 16 and 20 weeks (FACT-An Total and Cancer Linear Analogue Scale). Hb and Hematocrit levels were assessed at baseline, 4, 8, 12, 16 and 20 weeks. Transfusion requirements were recorded throughout the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Ortho Inc. Clinical Trial, Study Director — Janssen-Ortho Inc., Canada